CLINICAL TRIAL: NCT02193178
Title: Multicenter Dispensing Study of Biofinity Toric Made-To-Order Lenses in Extended Power Ranges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-14-05
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- comfilcon A toric (Experimental): Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
  Interventions: Device: comfilcon A Toric

INTERVENTIONS:
Device: comfilcon A Toric — Contact lenses
  Other Names: Biofinity

SUMMARY:
The study hypothesis is that the Biofinity Toric XR lenses will perform as well as or better than the participants' habitual contact lenses.

DETAILED DESCRIPTION:
The study hypothesis is that the Biofinity Toric XR lenses will perform as well as or better than the participants' habitual contact lenses. Further, that a minimum of 80% of those enrolled will complete 2 weeks of lens wear with no contraindication to continue.

ELIGIBILITY:
Inclusion Criteria:

* Has had an oculo-visual examination in the last two years
* Is at least 18 years of age and has full legal capacity to volunteer
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/50 or better (in at least one eye)
* Currently wears soft toric contact lenses in both eyes
* Subject contact lens prescription must fall under one of the contact lens power ranges for at least one eye:

  * -20.00D to -10.50D spherical powers and cylinder powers from - 0.75 to -2.25
  * +8.50D to +20.00D spherical powers and cylinder powers from - 0.75 to -2.25
  * -20.00D to -6.50D spherical powers and cylinder powers from -2.75 to -5.75
  * -6.00D to +6.00D spherical powers and cylinder powers from -2.75 to -5.75
  * +6.50D to +20.00D spherical powers and cylinder powers from-2.75 to -5.75
* Has clear corneas and no active ocular disease
* Demonstrates an acceptable fit with the study lenses

Exclusion Criteria:

* Has never worn contact lenses before;
* Has any systemic disease affecting ocular health;
* Is using any systemic or topical medications that will affect ocular health;
* Has any ocular pathology or abnormality that would affect the wearing of contact lenses;
* Has undergone corneal refractive surgery;
* Is participating in any other type of eye related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bergmanson, OD PhD, Principal Investigator — Texas Eye Research and Technology Center (TERTC), School of Optometry, University of Houston; Pete Kollbaum, OD PhD, Principal Investigator — Clinical Optics Research Lab (CORL), Indiana University School of Optometry, Indiana University
Locations (2):
- United States (2):
  - Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana
  - Texas Eye Research and Technology Center (TERTC) College of Optometry, University of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Period: Overall Study
Arm/Group | Overall Participants
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Dry eyes | 1

BASELINE CHARACTERISTICS:
Population: One participant discontinued and therefore data was not included in analysis.
Groups:
- Overall Baseline Characteristics: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Subjective ratings for overall comfort for habitual lenses assessed 2 weeks prior to baseline and for comfilcon A lenses assessed at baseline and 2 weeks post baseline. Scale 0-100, 0=cannot be worn, causes pain, and 100=cannot be felt ever.
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: One participant discontinued and therefore data was not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lenses; Comfilcon A - Baseline; Comfilcon A - 2 Weeks: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 14 | 13
units on a scale | 80 (16) | 91 (9) | 88 (11)

2. Primary Outcome: Overall Vision
Description: Subjective ratings for overall vision for habitual lenses assessed 2 weeks prior to baseline and vision for comfilcon A assessed at baseline and 2 weeks post.Scale 0-100, 0=Extremely poor vision all of the time, cannot function, 100=Excellent vision all of the time.
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post
Population: One participant discontinued and therefore data was not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 14 | 13
units on a scale | 75 (17) | 85 (15) | 80 (18)

3. Primary Outcome: Handling
Description: Subjective ratings for handling for habitual lenses assessed 2 weeks prior to baseline and handling for comfilcon A assessed at baseline and 2 weeks post baseline. Scale 0-100, 0=Very difficult, 100=Very easy
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: One participant discontinued and therefore data was not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 14 | 13
units on a scale | 88 (25) | 89 (16) | 94 (9)

4. Primary Outcome: Overall Satisfaction
Description: Subjective ratings for overall satisfaction for habitual lenses assessed 2 weeks prior to baseline and overall satisfaction for comfilcon A assessed at baseline and 2 weeks post baseline. Scale 0-100, 0=Extremely dissatisfied, 100=Extremely satisfied.
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: One participant discontinued and therefore data was not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 14 | 13
units on a scale | 90 (10) | 92 (9) | 89 (10)

5. Primary Outcome: Lens Fit - Rotation
Description: Lens Fit (rotation) for habitual lenses were assessed 2 weeks prior to baseline and then refitted with comfilcon A lenses. After refitting with comfilcon A, lens fit rotation was assessed at baseline and 2 weeks. Lens rotation was measured within 10 degrees of the desired 6 o'clock position. Scale 0-180 degrees, 0=no rotation, 180=max rotation.
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: One participant discontinued and therefore data was not included in analysis. Another participant did not wear habitual lens and therefore data was not collected for habitual lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 12 | 14 | 13
Number analyzed (eyes) | 24 | 28 | 26
percentage of eyes
  0 degrees | 18 | 29 | 21
  <=5 degrees | 64 | 71 | 64
  <=10 degrees | 93 | 86 | 89
  <=15 degrees | 93 | 93 | 93
  >15 degrees | 7 | 7 | 7

6. Primary Outcome: Lens Fit - Overall Stability
Description: Lens Fit (stability) for habitual lenses assessed 2 weeks prior to baseline and then refitted with comfilcon A lenses. After refitting with comfilcon A lenses, stability was assessed at baseline and 2 weeks. Scale 0-4, 0=Totally unstable, can't be worn to provide acceptable vision correction for an astigmatism, 4=Excellent orientation and optimum rotational recovery and stability
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Baseline; 2 Weeks: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Habitual Lenses | Baseline | 2 Weeks
Number analyzed (Participants) | 12 | 14 | 13
Number analyzed (eyes) | 24 | 28 | 26
units on a scale | 2.8 (0.7) | 3.3 (0.8) | 3.3 (0.6)

7. Primary Outcome: Lens Fit Acceptance
Description: General lens fit acceptance for habitual lenses assessed 2 weeks prior to baseline and refitted with comfilcon A lenses, which were assessed at baseline and at 2 weeks. (Scale 0-4, 0=Can't be worn; 4=Optimum)
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 12 | 14 | 13
Number analyzed (eyes) | 24 | 28 | 26
units on a scale | 3.0 (0.6) | 3.5 (0.7) | 3.3 (0.4)

8. Primary Outcome: Anterior Ocular Health - Palpebral Hyperemia and Roughness
Description: Palpebral hyperemia and roughness for comfilcon A lenses assessed at baseline and 2 weeks. Scale 0-4, 0=None, 4=Severe
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
Number analyzed (eyes) | 28 | 26
units on a scale
  Palpebral Conjunctival Hyperemia (Superior) | 0.75 (0.81) | 0.48 (0.33)
  Palpebral Conjunctival Hyperemia (Inferior) | 0.71 (0.60) | 0.50 (0.35)
  Palpebral Conjunctival Papillae (Superior) | 0.61 (0.46) | 0.58 (0.44)
  Palpebral Conjunctival Papillae (Inferior) | 0.64 (0.43) | 0.54 (0.37)

9. Primary Outcome: Anterior Ocular Health - Bulbar and Limbal Redness
Description: Bulbar and limbal redness for comfilcon A lenses assessed at baseline and 2 weeks. Scale 0-4, 0=None; 4=Severe injection
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
Number analyzed (eyes) | 28 | 26
units on a scale
  Bulbar (nasal) | 1.00 (0.71) | 0.67 (0.45)
  Bulbar (temporal) | 1.00 (0.75) | 0.67 (0.45)
  Bulbar (superior) | 0.79 (0.76) | 0.63 (0.46)
  Bulbar (inferior) | 0.79 (0.76) | 0.62 (0.45)
  Limbal (nasal) | 0.71 (1.07) | 0.21 (0.38)
  Limbal (temporal) | 0.71 (1.07) | 0.21 (0.38)
  Limbal (superior) | 0.80 (1.06) | 0.21 (0.38)
  Limbal (inferior) | 0.73 (1.09) | 0.19 (0.35)

10. Primary Outcome: Anterior Ocular Health - Corneal Staining
Description: Corneal staining for comfilcon A lenses assessed at baseline and 2 weeks. Scale 0-4, 0=No staining; 4= >45% of area
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
Number analyzed (eyes) | 28 | 26
units on a scale
  Central | 0.00 (0.00) | 0.00 (0.00)
  Nasal | 0.11 (0.31) | 0.04 (0.20)
  Temporal | 0.00 (0.00) | 0.00 (0.00)
  Superior | 0.04 (0.19) | 0.04 (0.20)
  Inferior | 0.11 (0.31) | 0.12 (0.33)

11. Primary Outcome: Anterior Ocular Health - Conjunctival Staining and Indentation
Description: Conjunctival staining and indentation for comfilcon A lenses assessed at baseline and 2 weeks. Conjuctival staining scale 0-4, 0=None, 4=Severe
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Conjunctival Staining (Baseline); Conjunctival Indentation (Baseline); Conjunctival Staining (2 Weeks); Conjunctival Indentation (2 Weeks): Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Conjunctival Staining (Baseline) | Conjunctival Indentation (Baseline) | Conjunctival Staining (2 Weeks) | Conjunctival Indentation (2 Weeks)
Number analyzed (Participants) | 14 | 14 | 13 | 13
Number analyzed (eyes) | 28 | 28 | 26 | 26
units on a scale
  Nasal | 0.34 (0.51) | 0.21 (0.40) | 0.54 (0.49) | 0.37 (0.52)
  Temporal | 0.23 (0.40) | 0.11 (0.31) | 0.29 (0.51) | 0.38 (0.50)
  Superior | 0.07 (0.18) | 0.00 (0.00) | 0.15 (0.31) | 0.02 (0.10)
  Inferior | 0.18 (0.43) | 0.13 (0.35) | 0.19 (0.38) | 0.21 (0.38)

12. Primary Outcome: Visual Acuity
Description: Visual acuity for habitual lenses assessed 2 weeks prior to baseline and for comfilcon A assessed at baseline and 2 weeks post baseline using logMAR.
Time Frame: 2 weeks prior to baseline, Baseline, 2 weeks post baseline
Population: One participant discontinued and therefore data was not included in analysis.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Habitual Lenses | Comfilcon A - Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 14 | 13
LogMAR
  High Contrast High Illumination (monocular) | 0.06 (0.14) | 0.06 (0.08) | 0.07 (0.14)
  High Contrast High Illumination (binocular) | -0.04 (0.09) | 0.00 (0.07) | -0.03 (0.09)
  High Contrast Low Illumination (monocular) | 0.19 (0.13) | 0.20 (0.09) | 0.23 (0.13)
  High Contrast Low Illumination (binocular) | 0.10 (0.09) | 0.15 (0.10) | 0.17 (0.14)

13. Primary Outcome: Subjective Preference - Comfort
Description: Subjective preference for comfort between habitual lenses and comfilcon A lenses assessed at baseline and 2 weeks. Preference choices: Prefers comfilcon A lenses, No preference, Prefers habitual lenses
Time Frame: Baseline and 2 weeks
Measure: Number; unit: percentage of subjects
Groups:
- Comfilcon A- Baseline; Comfilcon A-2 Weeks: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Comfilcon A- Baseline | Comfilcon A-2 Weeks
Number analyzed (Participants) | 14 | 13
percentage of subjects
  comfilcon A lenses | 57 | 69
  No preference | 43 | 23
  Habitual lenses | 0 | 8

14. Primary Outcome: Preference - Vision
Description: Subjective preference for vision between habitual lenses and comfilcon A lenses assessed at baseline and 2 weeks. Preference choices: Prefers comfilcon A lenses, No preference, Prefers habitual lenses
Time Frame: Baseline and 2 weeks
Measure: Number; unit: percentage of subjects
Groups:
- Comfilcon A Baseline; Comfilcon A - 2 Weeks: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Comfilcon A Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
percentage of subjects
  comfilcon A XR lenses | 50.0 | 46.2
  No preference | 28.6 | 15.4
  Habitual lenses | 21.4 | 38.5

15. Primary Outcome: Preference - Handling
Description: Subjective preference for handling between habitual lenses and comfilcon A lenses assessed at baseline and 2 weeks. Preference choices: Prefers comfilcon A lenses, No preference, Prefers habitual lenses
Time Frame: Baseline and 2 weeks
Population: Missing data for handling preference for one participant.
Measure: Number; unit: percentage of subjects
Arm/Group | Comfilcon A- Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
percentage of subjects
  comfilcon A lenses | 21.4 | 31
  No preference | 64.3 | 54
  Habitual lenses | 7.1 | 15
  Missing | 7.1 | 0

16. Primary Outcome: Overall Preference
Description: Overall subjective preference between habitual lenses and comfilcon A lenses assessed at baseline and 2 weeks. Preference choices: Prefers comfilcon A lenses, No preference, Prefers habitual lenses
Time Frame: Baseline and 2 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | Comfilcon A Baseline | Comfilcon A - 2 Weeks
Number analyzed (Participants) | 14 | 13
percentage of subjects
  comfilcon A lenses | 50 | 46
  No preference | 43 | 23
  Habitual lenses | 7 | 31

17. Primary Outcome: Investigator Acceptability
Description: Investigator's preference on acceptability of refitting subjects in to comfilcon A lens based on lens performance assessed at baseline and 2 weeks.Scale 1-5, 1=Strongly agree, 5=Strongly disagree.
Time Frame: Baseline and 2 weeks
Measure: Number; unit: percentage of subjects
Groups:
- Comfilcon A 2 Weeks: Participants are habitual toric lens wearers and will be fitted with comfilcon A toric lenses.
Arm/Group | Comfilcon A Baseline | Comfilcon A 2 Weeks
Number analyzed (Participants) | 14 | 13
percentage of subjects
  Agree | 86 | 85
  Neither Agree nor Disagree | 14 | 15
  Disagree | 0 | 0

ADVERSE EVENTS:
Time Frame: From dispense up to two weeks for each study lenses
Groups:
- Comfilcon A Toric XR MTO: Participants are habitual contact lens wearers and will be fitted with comfilcon A Toric XR MTO lenses.
  comfilcon A Toric XR (MTO) contact lenses
Arm/Group | Comfilcon A Toric XR MTO
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.